CLINICAL TRIAL: NCT01087229
Title: Comparative Study of the Effectiveness of an Equimolar Oxygen-nitrous Oxide Mixture During Physical Therapy for Adhesive Shoulder Capsulitis
Brief Title: Effectiveness of an Oxygen-nitrous Oxide Mixture During Physical Therapy for Frozen Shoulder
Acronym: MEOPA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHRC-I/2008/AD-01; 2008-007161-23 (EudraCT Number)
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Adhesive Capsulitis
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- equimolar oxygen-nitrous oxide mixture (Experimental): equimolar oxygen-nitrous oxide mixture
  Kinesitherapy is performed with a mask by which patient inhales an equimolar oxygen-nitrous oxide mixture.
  Interventions: Drug: equimolar oxygen-nitrous oxide mixture
- Placebo (Placebo Comparator): Patients randomized to this arm will have the placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: equimolar oxygen-nitrous oxide mixture — Kinesitherapy is performed with a mask by which patient inhales an equimolar oxygen-nitrous oxide mixture.
  Arms: equimolar oxygen-nitrous oxide mixture
Drug: Placebo — Kinesitherapy is performed with a mask by which patient inhales a placebo.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether or not the use of an equimolar mixture of oxygen and nitrous oxide during the physical therapy for patients suffering from frozen shoulder (adhesive shoulder capsulitis) results in a gain in shoulder amplitude (Constant Score) and less pain as compared to patients undergoing physical therapy without this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Affiliated with a social security system
* Has signed the consent form
* Patient has a painful, or initially painful but stable frozen shoulder (adhesive capsulitis): stiffening characterized by a passive loss of amplitude on three planes. This loss of amplitude is greater than or equal to 50% of controlateral amplitude when the controlateral shoulder is considered as normal. Otherwise, the loss of amplitude is greater than or equal to 50% of normal anatomical values.
* Radiography confirms the integrity of the glenohumeral interspace.

Exclusion Criteria:

* Intercurrent, evolving or unstable pathology: cancer, advanced cardio-vascular pathology, severe infection
* The patient is taking a treatment that may interfere with the study (eg corticoids, pain killers, chemotherapy)
* Contra-indication for physical therapy
* Coagulopathy
* Advanced diabetes mellitus, with neurological or joint complications
* Contra indication for the experimental treatment
* Pregnant or nursing women
* Patient's mental state prevents him/her from understanding the nature of the study, its objectives and potential consequences.
* Patient under guardianship
* Patient is in an exclusion period determined by a previous study
* Patient not able to follow protocol constraints or timetable
* Medical history of local infection, polyarthritis or neuropathy that might explain the shoulder pain.
* Absence of radiculopathy of cervical origin, of rotator cuff tears or evolving shoulder tendinopathy, of severe omarthrose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2010-03; Primary Completion 2013-09-02 (Actual); Study Completion 2013-09-02 (Actual)

PRIMARY OUTCOMES:
Change in the Constant Score using treatment as compared to without treatment. | fifteen days of physical therapy
  The Constant score questionnaire consists of 11 questions that result in a final score ranging from 0 to 100. The higher the test result, the more normally the shoulder is functioning.

SECONDARY OUTCOMES:
Change in kinetics at final session since baseline of passive glenohumeral flexion of the shoulder | Final session on Day 15
  Range of motion in degrees
Change in kinetics at final session since baseline of passive glenohumeral abduction of the shoulder | Final session on Day 15
  Range of motion in degrees
Change in kinetics at final session since baseline of passive glenohumeral external rotation (ER1) of the shoulder | Final session on Day 15
  Range of motion in degrees
Change in kinetics at final session since baseline of active global anterior flexion of the shoulder | Final session on Day 15
  Range of motion in degrees
Change in kinetics at final session since baseline of active global lateral flexion of the shoulder | Final session on Day 15
  Range of motion in degrees
Change in kinetics at final session since baseline of active global abduction of the shoulder | Final session on Day 15
  Range of motion in degrees
Change in kinetics at final session since baseline of active global external rotation (ER2) of the shoulder | Final session on Day 15
  Range of motion in degrees
Change in kinetics at final session since baseline of active global internal rotation of the shoulder | Final session on Day 15
  Range of motion in degrees
Change in kinetics at final session since baseline of passive global anterior flexion of the shoulder | Final session on Day 15
  Range of motion in degrees
Change in kinetics at final session since baseline of passive global lateral flexion of the shoulder | Final session on Day 15
  Range of motion in degrees
Change in kinetics at final session since baseline of passive global abduction of the shoulder | Final session on Day 15
  Range of motion in degrees
Change in kinetics at final session since baseline of passive global external rotation (ER2) of the shoulder | Final session on Day 15
  Range of motion in degrees
Pain at visits | At each session: final session on Day 15
  0-100 visual analogue scale (VAS)
Pain induced during sessions | At each session: final session on Day 15
  0-100 visual analogue scale (VAS)
Functional improvement | Day 7
  Disabilities of the Arm Shoulder and Hand scale (DASH)
Functional improvement | Day 15
  Disabilities of the Arm Shoulder and Hand scale (DASH)
Functional improvement | Day 45
  Disabilities of the Arm Shoulder and Hand scale (DASH)
Functional improvement | Day 180
  Disabilities of the Arm Shoulder and Hand scale (DASH)
Limitations posed to the physiotherapist activity due to patient pain at each session | At each session: final session on Day 15
  Likert six-point scale (none, to extremely high)
patient satisfaction | At each session: final session on Day 15
  0-10 VAS: 10=session interrupted due to pain; 0= session completed under perfect conditions
Change in the Constant Score using treatment as compared to without treatment | Day 7
Change in the Constant Score using treatment as compared to without treatment | Day 45
Change in the Constant Score using treatment as compared to without treatment | Day 180
Patient Quality of life | Day 1
  Medical Outcome Study Short Form-36 (MOS-SF36) score
Patient Quality of life | Day 7
  MOS-SF36 score
Patient Quality of life | Day 15
  MOS-SF36 score
Patient Quality of life | Day 45
  MOS-SF36 score
Patient Quality of life | Day 180
  MOS-SF36 score
Antalgic intake | Until end of study (Day 180)
  Discriptively noted

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Dupeyron, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (5):
- France (5):
  - Unité Rééducation Réadaptation Locomotrice, Le Grau-du-Roi, Gard
  - Centre Hospitalier Universitaire de Nîmes, Nîmes, Gard
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - CHU Lapeyronie, Montpellier
  - Centre Hélio Marin, Vallauris

REFERENCES:
- [Result] Dupeyron A, Dobija L, Castelli C, Petiot S, Tavares I, Gelis A, Coudeyre E. Nitrous oxide provided during intensive physiotherapy for shoulder adhesive capsulitis does not improve function: A randomised controlled trial. Ann Phys Rehabil Med. 2024 Apr;67(3):101803. doi: 10.1016/j.rehab.2023.101803. Epub 2023 Dec 19. PMID 38118247
- [Derived] Dupeyron A, Denarie M, Richard D, Dobija L, Castelli C, Petiot S, Tavares I, Gelis A, Coudeyre E. Analgesic gas for rehabilitation of frozen shoulder: Protocol for a randomized controlled trial. Ann Phys Rehabil Med. 2019 Jan;62(1):43-48. doi: 10.1016/j.rehab.2018.07.007. Epub 2018 Aug 9. PMID 30099150